CLINICAL TRIAL: NCT01070186
Title: Phase II, Open Label, Single Center Study of Sunitinib in Subjects With High Risk Renal Cell Carcinoma
Brief Title: Study of Sunitinib in Subjects With High Risk Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were enrolled.
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Fairooz Kabbinavar, MD / Principal Investigator, UCLA Jonsson Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-07-068
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Renal Cell Carcinoma
Keywords: nephrectomy; T1b; T2; T3; T4; N1; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sunitinib; Nephrectomy; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See intervention descriptions
  Interventions: Drug: Sunitinib; Other: Tumor biopsy; Procedure: Nephrectomy; Other: Biomarkers

INTERVENTIONS:
Drug: Sunitinib — 50mg/day for 4 weeks
  Other Names: Sutent
Other: Tumor biopsy — Conducted prior to administration of sunitinib therapy
Procedure: Nephrectomy — Nephrectomy 2-4 weeks after last dose of Sunitinib
Other: Biomarkers — Biomarker evaluation of blood prior to treatment, after 4 weeks of Sunitinib administration, and every three months for a year after surgery.
  Biomarker evaluation of tissue prior to 4 week administration of Sunitinib

SUMMARY:
This study is designed to explore the molecular modulatory effect of Sunitinib when given in a neoadjuvant setting prior to radical or partial nephrectomy. The study will evaluate aforementioned outcomes in 30 patients at a dose of 50mg/day for 4 weeks followed by surgery 2-4 weeks following the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Must be eligible to undergo a radical or partial nephrectomy
* Clinical stage T1b, T2, T3, T4 and/or N1 disease as documented by abdomen/pelvis CT scan, or MRI and chest x-ray or CT chest
* Patients must have a performance status on the ECOG scale of 0-1
* Patients must have a pretreatment wbc > 3.0, granulocyte count > 1000/mm3, hemoglobin > 8.5 g/dL, platelet count > 100,000/mm3 and a normal PT and PTT
* Patients must have a serum creatinine < 2.0 mg/dL
* Patients must have adequate hepatic function with a serum bilirubin < upper limit of normal and AST/ALT < 2.5 x upper limit of normal

Exclusion Criteria:

* Radiographic evidence of metastatic disease
* Prior administration of immunotherapy/biotherapy/hormonal or radiation for renal cell carcinoma
* Active secondary malignancies (other than basal cell carcinoma of the skin)
* Serious, nonhealing wound, ulcer, or bone fracture
* Clinically significant cardiovascular disease, New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication or Grade II or greater peripheral vascular disease within 1 year preceding Day 0
* Any history or radiologic evidence of central nervous system disease
* Active infection requiring parenteral antibiotics at the time of the first Sunitinib administration
* Current or recent (within the 10 days preceding Day 0) use of oral or parenteral anticoagulants (except as required to maintain patency of preexisting, permanency indwelling IV catheters), or aspirin
* Current, recent (within the 4 weeks preceding Day 0), or planned participation in another experimental drug study
* Screening clinical laboratory values:

  * ANC of < 1000/uL
  * Platelet count of < 100,000/uL
  * Total bilirubin > 2.0 mg/dL
  * AST or ALT > 2.5 times the upper limit of normal
  * Serum creatinine of > 2.0 mg/dL
  * Hemoglobin of < 9 gm/dL (may be transfused to maintain or exceed this level)
  * Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade > 2
  * Prolonged QTc interval on baseline EKG
  * Uncontrolled hypertension (>150/100 mm Hg despite optimal medical therapy)
  * Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
  * Patients receiving CYP3A4 inducers or inhibitors; patients should not take grapefruit juice or St. John's Wort while on the study
  * History of psychiatric disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
  * Unable to take medication by mouth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10

PRIMARY OUTCOMES:
Time to clinical recurrence after surgery for high risk localized disease. | 1 year

SECONDARY OUTCOMES:
Toxicity of Sunitinib when administered as neoadjuvant therapy prior to surgery | 1 year
  Toxicities will be graded using the NCI Common Toxicity Criteria, version 3.0
Effect of Sunitinib on pretreatment serum levels of Vascular Endothelial Growth Factor (VEGF). Tissue levels (biopsy and pathological specimen) of total VEGF, HIF-alpha, microvessel density, and apoptotic indices (TUNNEL Staining) | 1 year
Radiographically quantifiable evaluation of changes in cellular disorganization (marker of necrosis) and perfusion parameters before and during the administration of Sunitinib. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fairooz Kabbinavar, M.D., Principal Investigator — University of California, Los Angeles